CLINICAL TRIAL: NCT05633030
Title: Ureteral Access Sheath or Percutaneous Nephrostomy During Flexible Ureteroscopy: Which is Better?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, mohamed abdelrahman alhefnawy, assistant professor, Benha University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Ureteral access sheath or PCN
Record Dates: First submitted 2022-11-21; First posted 2022-12-01 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Flexible Ureteroscopy
Keywords: ureteral access sheath; ultrasound guided PCN

STUDY DESIGN:
Intervention Model Description: Group A: 50 patients will be operated using UAS during flexible ureteroscopy. Group B: 50 patients will be operated using PCN during flexible ureteroscopy.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- operated using UAS during flexible ureteroscopy (Active Comparator)
  Interventions: Procedure: using UAS during flexible ureteroscopy and using PCN during flexible ureteroscopy
- operated using PCN during flexible ureteroscopy (Active Comparator)
  Interventions: Procedure: using UAS during flexible ureteroscopy and using PCN during flexible ureteroscopy

INTERVENTIONS:
Procedure: using UAS during flexible ureteroscopy and using PCN during flexible ureteroscopy — under general anesthesia and given appropriate antibiotic cover. a clssic flexible ureteroscopy procedure is done and appropriately sized UAS was then inserted over the wire and positioned just distal to the PUJ or below upper ureteric stone under fluoroscopic guidance. We then perform a flexible ureteroscopy using Olympus URF-V2 (8.5 Fr) flexible ureteroscope to inspect the proximal ureter if there is upper ureteric stone, renal pelvis, and calyces for the presence of stones. Irrigation with 0.9% saline solution via a pressure-infusing system. Next, Holmium laser lithotripsy with a holmium:YAG laser [20 W; Lumenis (UK) Ltd., Elstree, UK] using a 272 micron laser fiber (Lumenis, Inc.) is carried out and/or stone extraction with a basket device, in the other group we add inserted trans papillary in the lower calyx of the kidney by an expert intervention radiologist

SUMMARY:
we aim to compare the safety and efficacy of flexible ureteroscopy with ureteral access sheath (group A) in comparison with flexible ureteroscopy without UAS but with PCN insertion (group B) either intra or post operaively by recording all data and the benefits , also comparing the drawbacks on each group

DETAILED DESCRIPTION:
A prospective randomized controlled study will be conducted at benha university hospitals on adult patients with renal and, or upper ureteric stones which will meet the inclusion criteria will participate in the study comparing usage of ureteral access sheath and percutaneous nephrostomy during flexible ureteroscopy. After filling out the informed consent form, patients will be randomly assigned to one of the two groups.

Group A: 50 patients will be operated using UAS during flexible ureteroscopy. Group B: 50 patients will be operated using PCN during flexible ureteroscopy.

Inclusion/Exclusion criteria:

Inclusion criteria consists of adult patients with upper ureteric stones and mild hydronephrosis or renal pelvic stones less than 20 mm with mild hydronephrosis.

Exclusion criteria include patients with active urinary tract infection and patients with uncontrolled coagulable status.

All patient demographics regarding age, gender, body mass index and comorbidities will be recorded. History, physical examination and laboratory investigations are done to exclude active urinary tract infection. Noncontrast computed tomography of the abdomen and plain abdominal radiography, so data revealed as stone side, stone burden, number of stones, hydronephrosis with its grade and Hounsfield Unit.

Technique

Group A: flexible ureteroscopy and UAS. Patients will be placed in the lithotomy position under general anesthesia and given appropriate antibiotic cover. The bladder and ureteric orifice will be directly visualized by rigid cystoscopy prior to the introduction of a safety guidewire., a semirigid ureteroscopy will be performed over a second working wire up to the pelvi-ureteric junction (PUJ) or as far proximally as safely achievable, allowing passive dilatation of the ureteric orifce and ureter. ureteral dilation using serial dilators is carried out if needed and up to 14 French (Fr). Two sizes of UAS were used: COOK Medical Flexor 12/14 French (Fr) (wider) and 9.5/11.5Fr (narrower). Appropriately sized UAS was then inserted over the wire and positioned just distal to the PUJ or below upper ureteric stone under fluoroscopic guidance. We then perform a flexible ureteroscopy using Olympus URF-V2 (8.5 Fr) flexible ureteroscope to inspect the proximal ureter if there is upper ureteric stone, renal pelvis, and calyces for the presence of stones. Irrigation with 0.9% saline solution via a pressure-infusing system. Next, Holmium laser lithotripsy with a holmium:YAG laser [20 W; Lumenis (UK) Ltd., Elstree, UK] using a 272 micron laser fiber (Lumenis, Inc.) is carried out and/or stone extraction with a basket device.

Group B: flexible ureteroscopy without UAS and insertion of PCN. Under general anesthesia in the supine position and given appropriate antibiotic, ultrasound guided 8 Fr PCN will be inserted trans papillary in the lower calyx of the kidney by an expert intervention radiologist. The bladder and ureteric orifice will be directly visualized by rigid cystoscopy prior to the introduction of a safety guidewire., a semi rigid ureteroscopy will be performed over a second working wire up to the pelviureteric junction (PUJ) or as far proximally as safely achievable, allowing passive dilatation of the ureteric orifice and ureter. ureteral dilation using serial dilators up to 10 Fr if needed. We then perform a flexible ureteroscopy using Olympus URF-V2 (8.5 Fr) flexible ureteroscope and complete procedure as described in the previous group and nephrostomy is open for irrigation and small dusted stone particles get its way out. At the end of the procedure, a double pigtail ureteral stent is left for 14 days. Once the operation is finished, PCN will be closed for 1 day and then the PCN catheter will be removed.

Operative time, intra-operative complications (bleeding, perforation, incompletion of procedure) and hospitalization periods will be recorded. Our follow-up protocol consisted of urinalysis, serum creatinine, and noncontrast computed tomography in the first month after the operation to assess stone-free rates and ureteral stricture formation, elevated serum creatinine level, and UTIs in the follow-up period. We will define success as the absence of any residual stones in the kidney or stone fragments less than 2 mm. Evaluation for success will be at 1 month and 3 months after the procedure.

Data management and analysis Quantitative data will be expressed as mean and standard deviation. Qualitative data will be expressed as frequencies and percent. Independent t-test will be used to assess the statistical significance of the difference between two study groups mean. Chi square test will be used to examine the relationship between qualitative data. The p <0.05 is considered significant in all tests. All statistics will be carried out using SPSS version 24 for Windows.

References

1. Donaldson JF, Lardas M, Scrimgeour D, Stewart F, MacLennan S, Lam TB, et al. Systematic review and meta-analysis of the clinical effectiveness of shock wave lithotripsy, retrograde intrarenal surgery, and percutaneous nephrolithotomy for lower-pole renal stones. Eur Urol. 2015;67:612-6.
2. Bozkurt OF, Resorlu B, Yildiz Y, Can CE, Unsal A. Retrograde intrarenal surgery versus percutaneous nephrolithotomy in the management of lower-pole renal stones with a diameter of 15 to 20 mm. J Endourol. 2011; 25:1131-5.
3. Pietrow PK, Auge BK, Delvecchio FC et al (2002) Techniques to maximize flexible ureteroscope longevity. Urology 60:784-788.
4. Gorin MA, Santos Cortes JA, Kyle CC et al (2015) Initial clinical experience with use of ureteral access sheaths in the diagnosis and treatment of upper tract urothelial carcinoma. Urology 78(3):523-527.
5. Guzelburc V, Guven S, Boz MY et al (2016) Intraoperative evaluation of ureteral access sheath-related injuries using post-ureteroscopic lesion scale. J Laparoendosc Adv Surg Tech A 26(1):23-26.
6. De Coninck, V.; Keller, E.X.; Rodriguez-Monsalve, M.; Audouin, M.; Doizi, S.; Traxer, O. Systematic review of ureteral access sheaths: Facts and myths. BJU Int. 2018, 122, 959-969.
7. Huang, J.; Zhao, Z.; AlSmadi, J.K.; Liang, X.; Zhong, F.; Zeng, T.; Wu, W.; Deng, T.; Lai, Y.; Liu, L.; et al. Use of the ureteral access sheath during ureteroscopy: A systematic review and meta-analysis. PLoS ONE 2018, 13, e0193600.
8. Traxer O, Thomas A (2013) Prospective evaluation and classification of ureteral wall injuries resulting from insertion of a ureteral access sheath during retrograde intrarenal surgery. J Urol 189:580-584.
9. Wright A, Williams K, Somani B et al (2015) Intrarenal pressure and irrigation flow with commonly used ureteric access sheaths and instruments. Cent Eur J Urol 68(4):434-438.
10. Goodwin WE, Casey WC, Woolf W. Percutaneous trocar (needle) nephrostomy in hydronephrosis. J Am Med Assoc 1955;157: 891-4.
11. Bell DA, Rose SC, Starr NK, Jaffe RB, Miller FJ Jr. Percutaneous nephrostomy for nonoperative management of fungal urinary tract infections. J Vasc Interv Radiol 1993;4:311-5
12. Mokhmalji H, Braun PM, Martinez Portillo FJ, Siegsmund M, Alken P, Kohrmann KU. Percutaneous nephrostomy versus ureteral stents for diversion of hydronephrosis caused by stones: a prospective, randomized clinical trial. J Urol 2001;165:1088-92
13. Lyncha MF, Ansona KM, Patelb U. Percutaneous nephrostomy and ureteric stent insertion for acute renal deobstruction consensus based guidance. J Clin Urol 2008;1:120-5.

ELIGIBILITY:
Inclusion Criteria:

* patients with upper ureteric stones and mild hydronephrosis or renal pelvic stones less than 20 mm with mild hydronephrosis

Exclusion Criteria:

* patients with active urinary tract infection and patients with uncontrolled coagulable status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
intra-operative complications | 3 mothes
  Operative time, intra-operative complications (bleeding, perforation, incompletion of procedure) and hospitalization periods

IPD SHARING:
Plan to Share IPD: Undecided